CLINICAL TRIAL: NCT03984812
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK3732394 in Healthy Participants
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics (PK) of GSK3732394 First-Time-in-Human (FTIH) Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early (following completion of SAD Cohort 3; 80 mg) based on PK/PD modelling which demonstrated the medicine's intended target profile was not achievable.
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207863
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: DAIDS, FTIH, HIV-1, MAD, SAD
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: In Part 1 of the study each of the subjects in the SAD cohorts (SAD Cohorts 1-5; SAD Cohort 6 is a possible expansion cohort that will be added as needed) will receive a single dose of blinded GSK3732394 or blinded PBO (GSK3732394: PBO = 6:2), per their randomization assignment. Part 2 will consist of up to three ascending repeat-dose cohorts (MAD Cohorts 1, 2, and 3), each with 8 subjects (blinded GSK3732394: blinded PBO = 6:2) will receive four weekly doses of GSK3732394 or PBO on Days 1, 8, 15, and 22.
Who Masked: Participant, Investigator
Masking Description: This is double-blind (sponsor-unblinded) study with subjects and the site staff blinded, except for an unblinded pharmacist at the site who will prepare the blinded drug product. The blind may be broken if, in the opinion of the investigator, it is in the subject's best interest for the investigator to know the study treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1,Cohort 1:Subjects receiving blinded GSK3732394 10mg/PBO (Experimental): GSK3732394 10 milligram (mg) or PBO will be administered by subcutaneous (SC) injection to the subjects.
  Interventions: Drug: GSK3732394; Drug: Placebo
- Part 1,Cohort 2:Subjects receiving blinded GSK3732394 40mg/PBO (Experimental): GSK3732394 40 mg or PBO will be administered by SC injection to the subjects. This is projected dose, dose will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3732394; Drug: Placebo
- Part1,Cohort 3:Subjects receiving blinded GSK3732394 130mg/PBO (Experimental): GSK3732394 130 mg or PBO will be administered by SC injection to the subjects. This is a projected dose. The dose administered in Part 1, Cohort 3 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3732394
- Part1,Cohort 4:Subjects receiving blinded GSK3732394 350mg/PBO (Experimental): GSK3732394 350 mg or PBO will be administered by SC injection to the subjects. This is a projected dose. The dose administered in Part 1, Cohort 4 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3732394; Drug: Placebo
- Part1,Cohort5: Subjects receiving blinded GSK3732394 600mg/PBO (Experimental): GSK3732394 600 mg or PBO will be administered by SC injection to the subjects. This is a projected dose. The dose administered in Part 1, Cohort 5 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3732394; Drug: Placebo
- Part1,Cohort6: Subjects receiving blinded GSK3732394 800mg/PBO (Experimental): GSK3732394 800 mg or PBO will be administered by SC injection to the subjects. This is a projected dose and will be given if necessary. The dose administered in Part 1, Cohort 6 (if necessary) will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3732394; Drug: Placebo
- Part2,Cohort1: Subjects receiving blinded GSK3732394 130mg/PBO (Experimental): GSK3732394 130 mg or PBO will be administered by SC injection to the subjects on Days 1, 8, 15, and 22 of the study. This is a projected dose. The dose administered in Part 2, Cohort 1 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3732394; Drug: Placebo
- Part2,Cohort2: Subjects receiving blinded GSK3732394 400mg/PBO (Experimental): GSK3732394 400 mg or PBO will be administered by SC injection to the subjects on Days 1, 8, 15, and 22 of the study. This is a projected dose. The administered dose in Part 2, Cohort 2 will be based on PK/PD results from preceding dosing cohorts.
  Interventions: Drug: GSK3732394; Drug: Placebo
- Part2,Cohort3: Subjects receiving blinded GSK3732394 600mg/PBO (Experimental): GSK3732394 600 mg or PBO will be administered by SC injection to the subjects on Days 1, 8, 15, and 22 of the study. This is a projected dose. The administered dose in Part 2, Cohort 3 will be based on PK/PD results from preceding dosing cohorts and will not exceed the maximum exposure observed in SAD (Part 1).
  Interventions: Drug: GSK3732394; Drug: Placebo

INTERVENTIONS:
Drug: GSK3732394 — It is composed of an anti-CD4 adnectin, an anti-N17 adnectin, and a peptide inhibitor. This will be provided as a solution for injection in 1 (milliliter) mL glass vials with the unit dose strength of 100 mg/mL
Drug: Placebo — Placebo will comprise of 0.9% weight per volume (w/v) sodium chloride.
  Arms: Part 1,Cohort 1:Subjects receiving blinded GSK3732394 10mg/PBO; Part 1,Cohort 2:Subjects receiving blinded GSK3732394 40mg/PBO; Part1,Cohort 4:Subjects receiving blinded GSK3732394 350mg/PBO; Part1,Cohort5: Subjects receiving blinded GSK3732394 600mg/PBO; Part1,Cohort6: Subjects receiving blinded GSK3732394 800mg/PBO; Part2,Cohort1: Subjects receiving blinded GSK3732394 130mg/PBO; Part2,Cohort2: Subjects receiving blinded GSK3732394 400mg/PBO; Part2,Cohort3: Subjects receiving blinded GSK3732394 600mg/PBO

SUMMARY:
This is a phase 1, 2-part, double-blind (sponsor-unblinded), randomized, placebo-controlled, FTIH study, that includes both single-ascending and multiple-ascending dose phase to assess the safety, tolerability, and pharmacokinetic (PK)/pharmacodynamic (PD) attributes of GSK3732394 in healthy subjects. The data gathered in this study will further enable clinical development of GSK3732394 in HIV-infected subjects. Approximately 72 healthy subjects will be randomized in the FTIH study. Part 1 will be the single ascending dose (SAD) phase and Part 2 will be the multiple ascending dose (MAD) phase. Each subject in the SAD cohort will receive a single dose of blinded GSK3732394 or blinded placebo (PBO) in 6:2 ratio. Part 1 will consist of five ascending single-dose cohorts with an additional expansion cohort included as needed. Part 2 will consist of up to three ascending repeat-dose cohorts (MAD Cohorts 1, 2, and 3), randomized to four weekly doses of blinded GSK3732394 or blinded PBO in 6:2 ratio to be administered on Days 1, 8, 15, and 22.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Subjects who are able to understand and comply with protocol requirements and timetables, instructions, and protocol-stated restrictions
* Body mass index within the range 19 to 30 kilogram per meter square (kg/m2) inclusive, in addition to a weight range of 50kg to 100kg.
* Male and female healthy volunteers.
* All male subjects must agree to use contraception during the treatment period and for at least 100 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies; Not a woman of childbearing potential (WOCBP), A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 28 days prior to first dose, and 40 days after, the last dose of study treatment.
* Capable of giving signed informed consent.
* A signed and dated written informed consent must be completed prior to the subject's entry into the study.

Exclusion Criteria:

* Subject has a history or presence of cardiovascular, dermatological, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Subject has abnormal blood pressure (as determined by the investigator).
* Subject had symptomatic herpes zoster within 3 months prior to screening.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, TB testing that includes a positive tuberculin skin test [TST]; defined as a skin induration greater than 5 millimeter [mm] at 48 to 72 hours,and regardless of Bacillus Calmette-Guerin [BCG] or other vaccination history) or a positive (not indeterminate) QuantiFERON-TB Gold test.
* Subjects with lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Subjects who had breast cancer within the past 10 years.
* Subjects who had history of severe injection site reaction (i.e., required emergency care or hospitalization) following any prior injection, including reaction to vaccines.
* Subjects with history of clinically significant allergy or prior hypersensitivity including those with a documented yeast allergy.
* Subjects with history of, or current concern for, a chronic immune deficiency disorder including, but not limited to: diabetes, sickle cell anemia, and malnutrition.
* Subjects having alanine transaminase (ALT) greater than 1.1 x upper limit of normal (ULN).
* Subjects with Hemoglobin levels below the normal range.
* Subjects with Platelet count <130,000 per cubic millimeters.
* Subjects with Creatinine clearance (CrCL) <90 milliliters per minute.
* Subjects with bilirubin greater than 1.1xULN (isolated bilirubin greater than 1.1xULN is acceptable if bilirubin is fractionated and direct bilirubin greater than 35%).
* Subjects who has current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects having Fridericia QT correction formula (QTcF) greater than 450 milliseconds (msec).
* Subjects who had intended use of over-the-counter or prescription medication within 7 days prior to dosing.
* Subjects who had live vaccine(s) within 1 month prior to screening, or plans to receive such vaccines during the study.
* Subjects who had treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Subjects who had exposure to immune-modulating medications (including corticosteroids) within 30-days of Screening.
* Subjects whose participation in the study would result in loss of blood or blood products in excess of 500 (milliliter) mL within 56 days.
* Subjects who had Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Subjects with current enrollment or past participation within the last 30 days before signing of consent in this or any other clinical study involving an investigational study intervention or any other type of medical research.
* Absolute CD4+ T-cell count and CD4 percent (CD4%) outside of the normal range for the reference laboratory (to be confirmed at baseline, e.g., Day -1).
* Subjects who had presence of Hepatitis B surface antigen (HBsAg) at screening.
* Subjects with positive Hepatitis C antibody test result at screening.
* Subjects with positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* Subjects with positive pre-study drug/alcohol screen.
* Subjects with positive human immunodeficiency virus (HIV) antibody test.
* Subjects with history of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 14 units. One unit is equivalent to 8 grams (g) of alcohol: a half pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Subjects with urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening.
* Subjects who has sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Krystal M, Chabria S, Austin D, Wolstenholme A, Wensel D, Lataillade M, Abberbock J, Baker M, Ackerman P. A Phase 1 randomized study of GSK3732394, an investigational long-acting biologic treatment regimen for HIV-1 infection. Antivir Ther. 2022 Oct;27(5):13596535221131164. doi: 10.1177/13596535221131164. PMID 36191080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was to have been a 2 part study, conducted to investigate single ascending doses (SAD) in Part 1 and repeated once-weekly multiple ascending doses (MAD) in Part 2. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Pre-assignment Details: A total of 24 healthy participants were enrolled in the study across the United States. This study was terminated due to non-safety reasons; hence, Part 1 (Cohorts 4 to 6) and Part 2 were not conducted.
Groups:
- Part 1- Cohort 1: GSK3732394 10 mg: Healthy adult participants were administered a single subcutaneous (SC) dose of blinded GSK3732394 10 milligrams (mg) on Day 1.
- Part 1- Cohort 2: GSK3732394 20 mg: Healthy adult participants were administered a single SC dose of blinded GSK3732394 20 mg on Day 1.
- Part 1- Cohort 3: GSK3732394 80 mg: Healthy adult participants were administered a single SC dose of blinded GSK3732394 80 mg on Day 1.
- Part 1- Placebo: Healthy adult participants were administered a single SC dose of blinded GSK3732394 matching placebo on Day 1 in cohorts 1, 2, and 3.
- Part 1- Cohort 4: GSK3732394; Part 1- Cohort 5: GSK3732394; Part 1- Cohort 6: GSK3732394: Healthy adult participants were planned to be administered a single SC dose of blinded GSK3732394
- Part 2- Cohort 1: GSK3732394; Part 2- Cohort 2: GSK3732394; Part 2- Cohort 3: GSK3732394: Healthy adult participants were planned to be administered a weekly dose of SC GSK3732394 on Days 1, 8, 15 and 22.
- Part 2: Placebo: Healthy adult participants were planned to be administered a weekly dose of SC GSK3732394 matching placebo on Days 1, 8, 15 and 22 in cohorts 1, 2 and 3.
Period: Part 1 (Up to Day 28)
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394 | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Started | 6 | 6 | 6 | 6 | 0 (No participants were enrolled in this arm as the study was terminated due to non-safety reasons.) | 0 (No participants were enrolled in this arm as the study was terminated due to non-safety reasons.) | 0 (No participants were enrolled in this arm as the study was terminated due to non-safety reasons.) | 0 | 0 | 0 | 0
Completed | 6 | 6 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Up to Day 49)
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394 | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (No participants were enrolled in Part 2 as the study was terminated due to non-safety reasons.) | 0 (No participants were enrolled in Part 2 as the study was terminated due to non-safety reasons.) | 0 (No participants were enrolled in Part 2 as the study was terminated due to non-safety reasons.) | 0 (No participants were enrolled in Part 2 as the study was terminated due to non-safety reasons.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only data for Part 1 is presented as study was terminated during Part 1; Part 2 was not initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394 | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] — Only data for Part 1 is presented as study was terminated during Part 1; Part 2 was not initiated.
  Years | 41.7 (5.82) | 34.3 (10.80) | 38.7 (6.95) | 33.0 (11.44) |  |  |  |  |  |  |  | 36.9 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Only data for Part 1 is presented as study was terminated during Part 1; Part 2 was not initiated.
  Participants
    Female | 1 | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Male | 5 | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Only data for Part 1 is presented as study was terminated during Part 1; Part 2 was not initiated.
  Participants
    African American/African Heritage | 2 | 1 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
    Asian- Japanese Heritage | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Asian- South East Asian Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    White- White/Caucasian/European Heritage | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
    American Indian/Alaskan Native and African American/African Heritage | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    American Indian/Alaskan Native and White/Caucasian/European Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Non-serious Adverse Event (SAEs) and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose: results in death and is life-threatening which requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity and birth defect or congenital anomaly, or any other situation that require medical or scientific judgement. Number of participants with common more than or equal to (>=)5 percent (%) non-serious AEs and SAEs are presented.
Time Frame: Up to Day 28
Population: Safety Population consisted of all participants who received at least 1 dose of study treatment. Participants will be analyzed according to the treatment they actually received. Data was not collected for Cohort 4 to 6, as the study was terminated after Part 1-Cohort 3 and hence no participants were enrolled. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants
  Non-SAEs | 4 | 4 | 4 | 2 |  |  |
  SAEs | 0 | 0 | 0 | 0 |  |  |

2. Primary Outcome: Part 2: Number of Participants With Non-SAEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose: results in death and is life-threatening which requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity and birth defect or congenital anomaly, or any other situation that require medical or scientific judgement. All AEs were planned to be collected from the start of treatment until the follow-up visit.
Time Frame: Up to Day 49
Population: Safety Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Clinical Chemistry Parameters by Maximum Grade Increase Post-Baseline
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: Glucose, alkaline phosphatase, alanine aminotransferase (ALT), amylase, aspartate aminotransferase (AST), direct bilirubin, total bilirubin, calcium, creatinine, potassium, lipase and sodium. The clinical chemistry abnormalities were graded using the Division of Acquired immunodeficiency syndrome (DAIDS) criteria and grades were derived based on numeric criteria as defined in DAIDS Version 2.1 and did not take into consideration of clinical signs or symptoms. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates more severe condition. Baseline is defined as the latest pre-dose assessment. Number of participants with clinical chemistry parameters by maximum grade increase post-Baseline is presented.
Time Frame: Up to Day 28
Population: Safety Population. Data was not collected for Cohort 4 to 6, as the study was terminated after Part 1-Cohort 3 and hence no participants were enrolled. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants
  Glucose; increase to Grade 1 | 0 | 0 | 1 | 0 |  |  |
  Glucose; increase to Grade 2 | 1 | 0 | 0 | 0 |  |  |
  Glucose; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Glucose; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Alkaline phosphatase; increase to Grade 1 | 0 | 0 | 0 | 0 |  |  |
  Alkaline phosphatase; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  Alkaline phosphatase; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Alkaline phosphatase; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  ALT, increase to Grade 1 | 0 | 0 | 0 | 0 |  |  |
  ALT, increase to Grade 2 | 1 | 0 | 0 | 0 |  |  |
  ALT, increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  ALT, increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Amylase; increase to Grade 1 | 1 | 1 | 1 | 1 |  |  |
  Amylase; increase to Grade 2 | 1 | 0 | 0 | 0 |  |  |
  Amylase; increase to Grade 3 | 0 | 0 | 0 | 1 |  |  |
  Amylase; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  AST; increase to Grade 1 | 1 | 1 | 0 | 2 |  |  |
  AST; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  AST; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  AST; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Direct bilirubin; increase to Grade 1 | 0 | 0 | 0 | 0 |  |  |
  Direct bilirubin; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  Direct bilirubin; increase to Grade 3 | 1 | 1 | 1 | 0 |  |  |
  Direct bilirubin; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Total bilirubin; increase to Grade 1 | 1 | 0 | 1 | 0 |  |  |
  Total bilirubin; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  Total bilirubin; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Total bilirubin; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Calcium; increase to Grade 1 | 1 | 2 | 0 | 0 |  |  |
  Calcium; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  Calcium; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Calcium; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Creatinine; increase to Grade 1 | 0 | 0 | 0 | 0 |  |  |
  Creatinine; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  Creatinine; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Creatinine; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Potassium; increase to Grade 1 | 1 | 0 | 0 | 0 |  |  |
  Potassium; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  Potassium; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Potassium; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Lipase: increase to Grade 1 | 1 | 0 | 0 | 1 |  |  |
  Lipase: increase to Grade 2 | 1 | 0 | 0 | 0 |  |  |
  Lipase: increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Lipase: increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |
  Sodium; increase to Grade 1 | 0 | 0 | 1 | 1 |  |  |
  Sodium; increase to Grade 2 | 0 | 0 | 0 | 0 |  |  |
  Sodium; increase to Grade 3 | 0 | 0 | 0 | 0 |  |  |
  Sodium; increase to Grade 4 | 0 | 0 | 0 | 0 |  |  |

4. Primary Outcome: Part 2: Number of Participants With Clinical Chemistry Parameters by Maximum Grade Increase Post-Baseline
Description: Blood samples were planned to be collected for the analysis of the following clinical chemistry parameters: Glucose, alkaline phosphatase, ALT, amylase, AST, direct and total bilirubin, calcium, creatinine, potassium, lipase and sodium. Baseline is defined as the latest pre-dose assessment.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Part 1: Number of Participants With Hematology Parameters by Maximum Grade Increase Post-Baseline
Description: Blood samples were collected for the analysis of following hematology parameters: Cluster of differentiation (CD) 4 cells, hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. The hematology abnormalities were graded using the DAIDS criteria and grades were derived based on numeric criteria as defined in DAIDS Version 2.1 and did not take into consideration of clinical signs or symptoms. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates more severe condition. Baseline is defined as the latest pre-dose assessment. Number of participants with hematology parameters by maximum grade increase post-Baseline is presented.
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants
  CD4; increase to grade 1 | 1 | 0 | 1 | 0 |  |  |
  CD4; increase to grade 2 | 0 | 0 | 0 | 0 |  |  |
  CD4; increase to grade 3 | 0 | 0 | 0 | 0 |  |  |
  CD4; increase to grade 4 | 0 | 0 | 0 | 0 |  |  |
  Hemoglobin; increase to grade 1 | 0 | 0 | 0 | 1 |  |  |
  Hemoglobin; increase to grade 2 | 0 | 0 | 0 | 0 |  |  |
  Hemoglobin; increase to grade 3 | 0 | 0 | 0 | 0 |  |  |
  Hemoglobin; increase to grade 4 | 0 | 0 | 0 | 0 |  |  |
  Lymphocytes; increase to grade 1 | 0 | 0 | 0 | 0 |  |  |
  Lymphocytes; increase to grade 2 | 0 | 0 | 0 | 0 |  |  |
  Lymphocytes; increase to grade 3 | 0 | 0 | 0 | 0 |  |  |
  Lymphocytes; increase to grade 4 | 0 | 0 | 0 | 0 |  |  |
  Neutrophils; increase to grade 1 | 0 | 0 | 0 | 0 |  |  |
  Neutrophils; increase to grade 2 | 0 | 0 | 0 | 0 |  |  |
  Neutrophils; increase to grade 3 | 0 | 0 | 0 | 0 |  |  |
  Neutrophils; increase to grade 4 | 0 | 0 | 0 | 0 |  |  |
  Platelets; increase to grade 1 | 0 | 0 | 0 | 0 |  |  |
  Platelets; increase to grade 2 | 0 | 0 | 0 | 0 |  |  |
  Platelets; increase to grade 3 | 0 | 0 | 0 | 0 |  |  |
  Platelets; increase to grade 4 | 0 | 0 | 0 | 0 |  |  |
  Leukocytes; increase to grade 1 | 0 | 0 | 0 | 0 |  |  |
  Leukocytes; increase to grade 2 | 0 | 0 | 0 | 0 |  |  |
  Leukocytes; increase to grade 3 | 0 | 0 | 0 | 0 |  |  |
  Leukocytes; increase to grade 4 | 0 | 0 | 0 | 0 |  |  |

6. Primary Outcome: Part 2: Number of Participants With Hematology Parameters by Maximum Grade Increase Post-Baseline
Description: Blood samples were planned to be collected for the analysis of the following hematology parameters: CD4 cells, hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. Baseline is defined as the latest pre-dose assessment.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Primary Outcome: Part 1: Number of Participants With Urinalysis Parameters by Any Increase in Discrete or Character Values Post Baseline
Description: Urine samples were collected for the analysis of urine parameters including bilirubin, glucose, ketones, leukocyte esterase, nitrite, occult blood, protein and urobilinogen. The urinalysis abnormalities were graded using the DAIDS criteria and grades were derived based on numeric criteria as defined in DAIDS Version 2.1 and did not take into consideration of clinical signs or symptoms. Baseline is defined as the latest pre-dose assessment. Number of participants with urinalysis parameters by any increase in discrete or character values post Baseline is presented.
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants
  Bilirubin; any increase | 0 | 0 | 0 | 0 |  |  |
  Glucose; any increase | 1 | 0 | 0 | 1 |  |  |
  Ketones; any increase | 1 | 0 | 1 | 2 |  |  |
  Leukocyte esterase; any increase | 0 | 2 | 1 | 3 |  |  |
  Nitrite; any increase | 0 | 0 | 0 | 2 |  |  |
  Occult blood; any increase | 4 | 4 | 3 | 2 |  |  |
  Protein; any increase | 1 | 1 | 1 | 1 |  |  |
  Urobilinogen; any increase; | 0 | 0 | 0 | 1 |  |  |

8. Primary Outcome: Part 2: Number of Participants With Urinalysis Parameters by Any Increase in Discrete or Character Values Post Baseline
Description: Urine samples were planned to be collected for the analysis of urine parameters including bilirubin, glucose, ketones, leukocyte esterase, nitrite, occult blood, protein and urobilinogen. Baseline is defined as the latest pre-dose assessment.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Primary Outcome: Part 1: Number of Participants With Worst Case Pulse Rate Post Baseline
Description: Pulse rate was measured in a semi-supine position after 5 minutes of rest. Participants are counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose value category are unchanged (e.g., High to High), or whose value became within range, are recorded in the "To within Range or No Change" category. Participants with missing Baseline value are assumed to have within range value. Participants were counted twice if the participant had both values that changed 'To Low' and 'To High'. Baseline is defined as the latest pre-dose assessment. Number of participants with pulse rate change to low or to high and no change post Baseline is presented.
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants
  To low | 0 | 0 | 0 | 0 |  |  |
  To high | 0 | 0 | 0 | 0 |  |  |
  No change | 6 | 6 | 6 | 6 |  |  |

10. Primary Outcome: Part 2: Number of Participants With Worst Case Pulse Rate Post Baseline
Description: Pulse rate was planned to be measured in a semi-supine position after 5 minutes of rest. Baseline is defined as the latest pre-dose assessment.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Primary Outcome: Part 1: Change From Baseline in Body Temperature
Description: Body temperature was measured in a semi-supine position after 5 minutes of rest. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and at Day 1 (1, 2, 4, 8, 12 hours), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: Safety Population. Data was not collected for Cohort 4 to 6, as the study was terminated after Part 1-Cohort 3 and hence no participants were enrolled. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles). Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Degrees Celsius
  Day 1: 1 hour; n= 6, 6, 6, 6, 0, 0, 0 | -0.08 (0.183) | 0.13 (0.216) | 0.00 (0.210) | -0.13 (0.361) |  |  |
  Day 1: 2 hours; n= 6, 6, 6, 6, 0, 0, 0 | -0.12 (0.417) | 0.08 (0.264) | 0.02 (0.117) | -0.05 (0.217) |  |  |
  Day 1: 4 hours; n= 6, 6, 6, 6, 0, 0, 0 | 0.02 (0.147) | 0.10 (0.110) | 0.08 (0.117) | 0.05 (0.226) |  |  |
  Day 1: 8 hours; n= 6, 6, 6, 6, 0, 0, 0 | -0.02 (0.098) | 0.13 (0.163) | 0.05 (0.152) | -0.10 (0.316) |  |  |
  Day 1: 12 hours; n= 6, 6, 6, 6, 0, 0, 0 | 0.00 (0.210) | 0.07 (0.175) | -0.02 (0.223) | -0.15 (0.164) |  |  |
  Day 2; n= 6, 6, 6, 6, 0, 0, 0 | -0.05 (0.217) | -0.05 (0.122) | -0.15 (0.084) | -0.17 (0.197) |  |  |
  Day 3; n = 6, 6, 6, 6, 0, 0, 0 | 0.08 (0.214) | 0.03 (0.163) | -0.12 (0.172) | -0.22 (0.214) |  |  |
  Day 4; n= 6, 6, 6, 6, 0, 0, 0 | 0.00 (0.200) | -0.03 (0.163) | -0.13 (0.344) | -0.08 (0.214) |  |  |
  Day 5; n= 6, 6, 6, 6, 0, 0, 0 | 0.03 (0.121) | 0.05 (0.197) | 0.03 (0.197) | -0.15 (0.138) |  |  |
  Day 6; n= 6, 6, 6, 6, 0, 0, 0 | -0.02 (0.183) | 0.00 (0.219) | -0.15 (0.327) | -0.05 (0.362) |  |  |
  Day 7; n= 6, 6, 6, 6, 0, 0, 0 | 0.03 (0.163) | 0.07 (0.207) | -0.02 (0.214) | 0.00 (0.155) |  |  |
  Day 8; n= 6, 6, 6, 6, 0, 0, 0 | -0.02 (0.160) | 0.00 (0.228) | 0.05 (0.235) | 0.00 (0.253) |  |  |
  Day 9; n= 6, 6, 6, 6, 0, 0, 0 | -0.02 (0.160) | -0.08 (0.232) | -0.05 (0.315) | -0.10 (0.167) |  |  |
  Day 10; n= 6, 6, 6, 6, 0, 0, 0 | 0.03 (0.121) | -0.07 (0.175) | 0.05 (0.327) | -0.03 (0.151) |  |  |
  Day 11; n= 6, 6, 6, 6, 0, 0, 0 | 0.07 (0.137) | 0.07 (0.266) | -0.15 (0.187) | -0.12 (0.204) |  |  |
  Day 12; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  Day 12; n= 6, 5, 6, 6, 0, 0, 0 | -0.05 (0.274) | -0.02 (0.130) | -0.02 (0.117) | -0.03 (0.234) |  |  |
  Day 13; n= 6, 6, 6, 6, 0, 0, 0 | 0.02 (0.172) | 0.05 (0.197) | -0.02 (0.271) | -0.05 (0.259) |  |  |
  Day 14; n= 6, 6, 6, 6, 0, 0, 0 | 0.08 (0.172) | 0.03 (0.356) | -0.08 (0.172) | 0.02 (0.117) |  |  |
  Day 17; n= 6, 6, 6, 6, 0, 0, 0 | 0.10 (0.179) | -0.17 (0.437) | -0.05 (0.187) | -0.13 (0.151) |  |  |
  Day 21; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  Day 21; n= 6, 5, 6, 6, 0, 0, 0 | 0.00 (0.110) | 0.06 (0.195) | -0.05 (0.295) | -0.23 (0.273) |  |  |
  Day 24; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  Day 24; n= 6, 5, 6, 6, 0, 0, 0 | -0.03 (0.121) | 0.22 (0.295) | -0.08 (0.306) | -0.12 (0.240) |  |  |
  Day 28; n= 6, 6, 6, 6, 0, 0, 0 | 0.10 (0.167) | 0.03 (0.308) | 0.10 (0.253) | -0.15 (0.295) |  |  |

12. Primary Outcome: Part 2: Change From Baseline in Body Temperature
Description: Body temperature was planned to be measured in a semi-supine position after 5 minutes of rest. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Primary Outcome: Part 1: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in a semi-supine position after 5 minutes of rest. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and at Day 1 (1, 2, 4, 8, 12 hours), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Breaths per minute
  Day 1: 1 hour; n= 6, 6, 6, 6, 0, 0, 0 | -0.2 (2.23) | 0.0 (2.53) | -0.3 (2.25) | 0.2 (2.04) |  |  |
  Day 1: 2 hours; n= 6, 6, 6, 6, 0, 0, 0 | 0.0 (2.19) | 2.7 (1.63) | 0.0 (1.26) | 0.0 (1.79) |  |  |
  Day 1: 4 hours; n= 6, 6, 6, 6, 0, 0, 0 | 0.0 (3.35) | 0.0 (1.79) | -2.8 (2.56) | 0.0 (2.83) |  |  |
  Day 1: 8 hours; n= 6, 6, 6, 6, 0, 0, 0 | 2.7 (2.94) | 0.0 (1.79) | -0.3 (3.44) | -0.3 (2.66) |  |  |
  Day 1: 12 hours; n= 6, 6, 6, 6, 0, 0, 0 | 2.2 (2.71) | 2.2 (2.32) | 1.0 (2.19) | 2.0 (3.58) |  |  |
  Day 2; n= 6, 6, 6, 6, 0, 0, 0 | -0.3 (3.14) | 0.8 (2.71) | -0.5 (1.22) | 1.3 (2.42) |  |  |
  Day 3; n = 6, 6, 6, 6, 0, 0, 0 | 0.0 (3.10) | 0.7 (2.73) | -1.8 (2.71) | 0.0 (3.35) |  |  |
  Day 4; n= 6, 6, 6, 6, 0, 0, 0 | 0.0 (4.00) | -1.3 (1.63) | -2.2 (1.83) | -0.7 (2.07) |  |  |
  Day 5; n= 6, 6, 6, 6, 0, 0, 0 | 1.3 (2.42) | 0.7 (2.07) | 0.2 (2.40) | 0.7 (1.63) |  |  |
  Day 6; n= 6, 6, 6, 6, 0, 0, 0 | -0.3 (2.66) | 1.3 (1.63) | -1.5 (2.51) | 2.3 (1.97) |  |  |
  Day 7; n= 6, 6, 6, 6, 0, 0, 0 | -1.2 (2.99) | 0.2 (1.33) | -2.3 (3.39) | -1.3 (1.63) |  |  |
  Day 8; n= 6, 6, 6, 6, 0, 0, 0 | 1.3 (1.03) | 1.3 (2.73) | -0.2 (2.04) | 0.5 (2.66) |  |  |
  Day 9; n= 6, 6, 6, 6, 0, 0, 0 | -1.0 (3.35) | -0.3 (3.67) | 0.5 (1.97) | 0.5 (1.52) |  |  |
  Day 10; n= 6, 6, 6, 6, 0, 0, 0 | -0.3 (2.66) | 1.3 (2.42) | -0.5 (2.66) | 1.3 (3.27) |  |  |
  Day 11; n= 6, 6, 6, 6, 0, 0, 0 | -0.3 (3.20) | -1.3 (2.07) | -1.5 (3.45) | 0.7 (3.72) |  |  |
  Day 12; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  Day 12; n= 6, 5, 6, 6, 0, 0, 0 | 0.0 (2.19) | 0.4 (2.61) | -0.8 (2.23) | 0.5 (2.35) |  |  |
  Day 13; n= 6, 6, 6, 6, 0, 0, 0 | -2.0 (3.10) | -1.7 (2.34) | -0.2 (1.60) | 0.3 (4.46) |  |  |
  Day 14; n= 6, 6, 6, 6, 0, 0, 0 | 0.3 (1.97) | 0.7 (1.03) | -0.2 (1.83) | 0.3 (1.51) |  |  |
  Day 17; n= 6, 6, 6, 6, 0, 0, 0 | 1.0 (1.67) | 1.0 (1.67) | 0.5 (2.51) | 1.2 (2.40) |  |  |
  Day 21; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  Day 21; n= 6, 5, 6, 6, 0, 0, 0 | 0.3 (2.34) | 1.2 (2.28) | 1.0 (1.55) | 0.0 (1.79) |  |  |
  Day 24; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  Day 24; n= 6, 5, 6, 6, 0, 0, 0 | 1.3 (1.63) | 0.2 (2.28) | -0.5 (1.22) | 1.0 (1.67) |  |  |
  Day 28; n= 6, 6, 6, 6, 0, 0, 0 | -0.7 (3.01) | 1.7 (1.51) | -0.2 (2.56) | 1.0 (1.10) |  |  |

14. Primary Outcome: Part 2: Change From Baseline in Respiratory Rate
Description: Respiratory rate was planned to be measured in a semi-supine position after 5 minutes of rest. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Primary Outcome: Part 1: Number of Participants With Worst Case Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Post Baseline
Description: SBP and DBP was measured in a semi-supine position after 5 minutes of rest. Participants are counted in the worst case category that their value changes to low, within range or no change, or high), unless there is no change in their category. Participants whose value category are unchanged (e.g., High to High), or whose value became within range, are recorded in the "To within Range or No Change" category. Participants with missing Baseline value are assumed to have within range value. Participants were counted twice if the participant had both values that changed 'To Low' and 'To High'. Baseline is defined as the latest pre-dose assessment. Number of participants with SBP and DBP change to low and to high and no change post Baseline is presented.
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants
  SBP: To low | 0 | 0 | 0 | 0 |  |  |
  SBP: To high | 0 | 0 | 0 | 0 |  |  |
  SBP: No change | 6 | 6 | 6 | 6 |  |  |
  DBP: To low | 0 | 0 | 1 | 0 |  |  |
  DBP: To high | 0 | 0 | 0 | 0 |  |  |
  DBP: No change | 6 | 6 | 5 | 6 |  |  |

16. Primary Outcome: Part 2: Number of Participants With Worst Case SBP and DBP Post Baseline
Description: SBP and DBP was planned to be measured in a semi-supine position after 5 minutes of rest. Baseline is defined as the latest pre-dose assessment.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Primary Outcome: Part 1: Number of Participants With Clinical Significant Abnormal Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of 5 minutes. Twelve lead ECGs were obtained by using an automated ECG machine. Number of participants with clinical significant abnormal ECG findings are presented.
Time Frame: Pre-dose, 4, 12 hours on Day 1, 24 hours on Day 2, Days 8, 14, 17 and 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants
  Day 1- Pre-dose | 0 | 0 | 0 | 0 |  |  |
  Day 1- 4 hours | 0 | 0 | 0 | 0 |  |  |
  Day 1- 12 hours | 0 | 0 | 0 | 0 |  |  |
  Day 2- 24 hours | 0 | 0 | 0 | 0 |  |  |
  Day 8 | 0 | 0 | 0 | 0 |  |  |
  Day 14 | 0 | 0 | 0 | 0 |  |  |
  Day 17 | 0 | 0 | 0 | 0 |  |  |
  Day 28 | 0 | 0 | 0 | 0 |  |  |

18. Primary Outcome: Part 2: Number of Participants With Clinical Significant Abnormal ECG Findings
Description: 12-lead ECG recordings was planned to be measured.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Part 1: Area Under the Plasma Concentration Time Curve From Zero to t (AUC[0-t]) Following Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3732394. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: PK Population consisted of all participants in the Safety population who had at least 1 non-missing PK assessment. Data was not collected for Cohort 4 to 6, as the study was terminated after Part 1-Cohort 3 and hence no participants were enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Hours*micrograms per milliliter | 10.904 (152.1) | 26.823 (69.1) | 111.065 (42.1) |  |  |

20. Secondary Outcome: Part 2: AUC(0-t) After Repeat Dosing of GSK3732394 in First Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6 and 7
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-infinity]) Following Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for PK analysis of GSK3732394. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: PK Population. Data was not collected for Cohort 4 to 6, as the study was terminated after Part 1-Cohort 3 and hence no participants were enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Hours*micrograms per milliliter | 18.414 (50.4) | 28.242 (66.4) | 112.215 (41.7) |  |  |

22. Secondary Outcome: Part 2: AUC(0-infinity) After Repeat Dosing of GSK3732394 in First Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6 and 7
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) Following Single Dose Administration of GSK3732394
Description: as for outcome 21
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Micrograms per milliliter | 0.18376 (130.5) | 0.38693 (81.3) | 1.25024 (49.7) |  |  |

24. Secondary Outcome: Part 2: Cmax After Repeat Dosing of GSK3732394 in First Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6 and 7
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Part 2: Cmax After Repeat Dosing of GSK3732394 in Last Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Part 1: Time of Occurrence of Cmax (Tmax) After Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for PK analysis of GSK3732394. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Hours | 24.0 [12 to 48] | 24.0 [12 to 48] | 48.0 [24 to 72] |  |  |

27. Secondary Outcome: Part 2: Tmax After Repeat Dosing of GSK3732394 in First Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6 and 7
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Part 2: Tmax After Repeat Dosing of GSK3732394 in Last Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: Part 1: Lag Time Before Observation of Drug Concentrations (Tlag) After Single Dose Administration of GSK3732394
Description: as for outcome 26
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Hours | 3.00 [1.0 to 12.0] | 1.50 [1.0 to 2.0] | 1.50 [0.5 to 2.0] |  |  |

30. Secondary Outcome: Part 2: Tlag After Repeat Dosing of GSK3732394 in First Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6 and 7
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Part 1: Last Observable Concentration (Clast) After Single Dose Administration of GSK3732394
Description: as for outcome 21
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Micrograms per milliliter | 0.03974 (34.0) | 0.03528 (27.2) | 0.03245 (21.8) |  |  |

32. Secondary Outcome: Part 1: Time of Last Observable Concentration (Tlast) After Single Dose Administration of GSK3732394
Description: as for outcome 21
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Hours | 96.0 [72 to 144] | 132.0 [120 to 168] | 192.0 [192 to 216] |  |  |

33. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (t1/2) After Single Dose Administration of GSK3732394
Description: as for outcome 21
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Hours | 27.326 [23.78 to 36.43] | 25.084 [19.33 to 27.79] | 22.517 [17.44 to 28.55] |  |  |

34. Secondary Outcome: Part 2: T1/2 After Repeat Dosing of GSK3732394 in Last Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Part 1: Apparent Clearance (CL/F) After Single Dose Administration of GSK3732394
Description: as for outcome 21
Time Frame: Day 1 (Pre-dose, 0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0
Liters per hour | 0.543 (50.4) | 0.708 (66.4) | 0.713 (41.7) |  |  |

36. Secondary Outcome: Part 2: CL/F After Repeat Dosing of GSK3732394 in Last Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

37. Secondary Outcome: Part 2: Area Under the Concentration Time Curve at Steady State Within the Dosing Interval (AUC[0-tau]) After Repeat Dosing of GSK3732394 in Last Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Part 2: Trough Concentration (Ctrough) After Repeat Dosing of GSK3732394 in Last Week
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394.
Time Frame: Day 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

39. Secondary Outcome: Part 2: Accumulation Ratio Using AUC(0-tau) (RAUC[0-tau]) After Repeat Dosing of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394. RAUC(0-tau) was planned to be calculated as the ratio of AUC(0-tau) on week 4 to AUC(0-tau) on week 1 .
Time Frame: Days 1 and 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6, 7, 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

40. Secondary Outcome: Part 2: Accumulation Ratio Using Cmax (RCmax) After Repeat Dosing of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394. RCmax was planned to be calculated as the ratio of Cmax on Week 4 to Cmax on Week 1.
Time Frame: Days 1 and 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6, 7, 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

41. Secondary Outcome: Part 2: Accumulation Ratio Using Ctrough (RCtrough) After Repeat Dosing of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3732394. RCtrough was planned to be calculated as the ratio of Ctrough on Week 4 to Ctrough on Week 1.
Time Frame: Days 1 and 22 (pre-dose, 0.5, 1, 2, 4, 8 and 12 hours), Days 2, 3, 4, 5, 6, 7, 23, 24, 25, 26, 27 and 28
Population: PK Population. Data was not collected for Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394
Number analyzed (Participants) | 0 | 0 | 0

42. Secondary Outcome: Part 1: Change From Baseline in Percent of CD4 Receptor Occupancy (RO) After Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for Pharmacodynamic (PD) analysis of CD4 receptors occupied by GSK3732394 on CD4+ T cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline, Day 1 (0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage of CD4 receptor occupancy
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Percentage of CD4 receptor occupancy
  %CD4 RO; Day 1- 0.5 hours; n= 6, 6, 6, 6, 0, 0, 0 | -1.05 (3.237) | -0.55 (2.723) | -4.25 (8.090) | -5.27 (18.843) |  |  |
  %CD4 RO; Day 1- 1 hour; n= 6, 6, 6, 6, 0, 0, 0 | -2.67 (4.141) | -0.60 (4.995) | -2.57 (6.038) | -8.95 (19.146) |  |  |
  %CD4 RO; Day 1- 2 hours; n= 6, 6, 6, 6, 0, 0, 0 | -2.23 (8.023) | -1.00 (6.078) | 1.10 (5.277) | -5.78 (15.581) |  |  |
  %CD4 RO; Day 1- 4 hours; n= 6, 6, 6, 6, 0, 0, 0 | -0.03 (3.355) | 1.38 (5.401) | 3.27 (11.005) | -5.37 (21.701) |  |  |
  %CD4 RO; Day 1- 8 hours; n= 6, 6, 6, 6, 0, 0, 0 | -6.72 (5.689) | -1.85 (20.766) | 15.03 (14.890) | -12.27 (23.916) |  |  |
  %CD4 RO; Day 1- 12 hours; n= 6, 6, 6, 6, 0, 0, 0 | -8.13 (8.504) | -2.28 (15.546) | 14.43 (18.026) | -11.20 (22.067) |  |  |
  %CD4 RO; Day 2; n= 6, 6, 6, 6, 0, 0, 0 | -4.02 (8.737) | 3.58 (25.018) | 33.12 (20.937) | -9.62 (25.708) |  |  |
  %CD4 RO; Day 3; n= 6, 6, 6, 6, 0, 0, 0 | 5.35 (6.954) | 10.53 (21.504) | 32.63 (16.428) | -10.30 (15.514) |  |  |
  %CD4 RO; Day 4; n= 6, 6, 6, 6, 0, 0, 0 | -4.80 (20.651) | 12.13 (15.666) | 27.72 (16.784) | -10.70 (13.301) |  |  |
  %CD4 RO; Day 5; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  %CD4 RO; Day 5; n= 6, 5, 6, 6, 0, 0, 0 | -5.28 (9.691) | -2.56 (25.413) | 23.75 (17.113) | -17.57 (19.174) |  |  |
  %CD4 RO; Day 6; n= 6, 6, 6, 6, 0, 0, 0 | -4.03 (9.002) | -0.12 (10.732) | 17.97 (10.318) | -15.82 (18.704) |  |  |
  %CD4 RO; Day 7; n= 6, 6, 6, 6, 0, 0, 0 | -12.77 (9.550) | -12.63 (10.287) | 11.13 (13.077) | -13.13 (14.586) |  |  |
  %CD4 RO; Day 8; n= 6, 6, 6, 6, 0, 0, 0 | -5.93 (15.457) | -14.62 (7.440) | 10.92 (12.357) | -17.38 (16.299) |  |  |
  %CD4 RO; Day 9; n= 6, 6, 6, 6, 0, 0, 0 | -7.90 (5.197) | -15.40 (6.874) | 6.47 (9.276) | -16.12 (23.008) |  |  |
  %CD4 RO; Day 10; n= 6, 6, 6, 6, 0, 0, 0 | -6.25 (4.127) | -23.55 (11.248) | 1.70 (14.214) | -16.55 (26.904) |  |  |
  %CD4 RO; Day 11; n= 6, 6, 6, 6, 0, 0, 0 | -8.53 (10.003) | -15.57 (6.905) | -0.55 (6.568) | -12.50 (16.236) |  |  |
  %CD4 RO; Day 12; n= 5, 6, 6, 6, 0, 0, 0: number analyzed (Participants) | 5 | 6 | 6 | 6 | 0 | 0 | 0
  %CD4 RO; Day 12; n= 5, 6, 6, 6, 0, 0, 0 | -6.94 (8.481) | -20.12 (8.206) | -4.83 (6.508) | -19.17 (17.995) |  |  |
  %CD4 RO; Day 13; n= 6, 6, 6, 6, 0, 0, 0 | -8.98 (4.830) | -17.40 (3.347) | -5.00 (7.812) | -19.75 (28.071) |  |  |
  %CD4 RO; Day 14; n= 6, 6, 6, 5, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0 | 0
  %CD4 RO; Day 14; n= 6, 6, 6, 5, 0, 0, 0 | -11.35 (10.882) | -21.40 (7.461) | -9.40 (4.268) | -20.10 (8.317) |  |  |
  %CD4 RO; Day 17; n= 6, 6, 6, 6, 0, 0, 0 | -7.45 (5.767) | -20.28 (8.181) | -7.47 (12.876) | -10.42 (11.522) |  |  |
  %CD4 RO; Day 21; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  %CD4 RO; Day 21; n= 6, 5, 6, 6, 0, 0, 0 | -14.18 (6.563) | -21.00 (11.299) | -5.47 (12.620) | -12.98 (21.314) |  |  |
  %CD4 RO; Day 24; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  %CD4 RO; Day 24; n= 6, 5, 6, 6, 0, 0, 0 | -18.75 (7.908) | -23.32 (4.751) | -7.62 (6.751) | -17.22 (23.678) |  |  |
  %CD4 RO; Day 28; n= 6, 6, 6, 6, 0, 0, 0 | -12.20 (7.215) | -18.35 (6.778) | -10.17 (6.532) | -22.95 (25.642) |  |  |

43. Secondary Outcome: Part 2: Change From Baseline in Percent of CD4 RO After Multiple Dose Administration of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for PD analysis of CD4 receptors occupied by GSK3732394 on CD4+ T cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

44. Secondary Outcome: Part 1: Change From Baseline in CD3+ Cells Following Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for analysis of CD3+ cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline, Days 2, 3, 5, 8, 11, 14, 17, 21, 24 and 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
10^9 cells per Liter
  CD3+; Day 2;n= 6, 6, 6, 6, 0, 0, 0 | -0.1062 (0.11203) | -0.1770 (0.21913) | -0.1250 (0.15424) | -0.2353 (0.18327) |  |  |
  CD3+: Day 3; n= 6, 6, 6, 6, 0, 0, 0 | -0.1655 (0.21564) | -0.0582 (0.18274) | -0.2420 (0.18457) | -0.1862 (0.12896) |  |  |
  CD3+: Day 5; n= 6, 6, 5, 6, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0 | 0 | 0
  CD3+: Day 5; n= 6, 6, 5, 6, 0, 0, 0 | -0.1653 (0.16295) | -0.1963 (0.12555) | -0.1884 (0.24561) | -0.2713 (0.14030) |  |  |
  CD3+; Day 8; n= 6, 6, 6, 6, 0, 0, 0 | -0.1490 (0.17208) | -0.1418 (0.22769) | -0.2110 (0.22989) | -0.1548 (0.07763) |  |  |
  CD3+; Day 11; n= 6, 6, 6, 6, 0, 0, 0 | -0.1152 (0.11569) | -0.2120 (0.25092) | -0.1760 (0.20947) | -0.2410 (0.18211) |  |  |
  CD3+; Day 14; n= 6, 6, 6, 5, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0 | 0
  CD3+; Day 14; n= 6, 6, 6, 5, 0, 0, 0 | -0.1735 (0.29145) | -0.3187 (0.26375) | -0.2372 (0.19635) | -0.2326 (0.15181) |  |  |
  CD3+; Day 17; n= 6, 6, 6, 6, 0, 0, 0 | -0.1412 (0.21510) | -0.1302 (0.29482) | -0.0215 (0.34581) | -0.1647 (0.11501) |  |  |
  CD3+; Day 21; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD3+; Day 21; n= 6, 5, 6, 6, 0, 0, 0 | -0.0823 (0.12965) | -0.2802 (0.31982) | -0.0958 (0.35546) | -0.2733 (0.12373) |  |  |
  CD3+; Day 24; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD3+; Day 24; n= 6, 5, 6, 6, 0, 0, 0 | -0.1448 (0.27643) | -0.3532 (0.19601) | -0.1790 (0.35340) | -0.3267 (0.20015) |  |  |
  CD3+; Day 28; n= 6, 6, 6, 6, 0, 0, 0 | -0.1047 (0.17612) | -0.0273 (0.32856) | -0.3340 (0.20039) | -0.2688 (0.26645) |  |  |

45. Secondary Outcome: Part 2: Change From Baseline in CD3+ Cells Following Multiple Dose Administration of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for analysis of CD3+ cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

46. Secondary Outcome: Part 1: Change From Baseline in CD4+ Cells Following Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for analysis of CD4+ cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline, Days 2, 3, 5, 8, 11, 14, 17, 21, 24 and 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^6 cells per Liter
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
10^6 cells per Liter
  CD4+; Day 2;n= 6, 6, 6, 6, 0, 0, 0 | -38.2 (45.39) | -150.2 (161.86) | -82.0 (88.85) | -128.5 (104.57) |  |  |
  CD4+: Day 3; n= 6, 6, 6, 6, 0, 0, 0 | -84.3 (98.77) | -55.8 (125.97) | -158.0 (95.88) | -94.0 (79.39) |  |  |
  CD4+: Day 5; n= 6, 6, 5, 6, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0 | 0 | 0
  CD4+: Day 5; n= 6, 6, 5, 6, 0, 0, 0 | -72.5 (71.47) | -138.8 (98.39) | -142.2 (166.65) | -159.0 (72.39) |  |  |
  CD4+; Day 8; n= 6, 6, 6, 6, 0, 0, 0 | -78.5 (105.58) | -108.5 (173.59) | -133.0 (165.72) | -89.2 (80.55) |  |  |
  CD4+; Day 11; n= 6, 6, 6, 6, 0, 0, 0 | -63.5 (63.52) | -159.2 (169.61) | -126.0 (168.61) | -136.7 (136.59) |  |  |
  CD4+; Day 14; n= 6, 6, 6, 5, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0 | 0
  CD4+; Day 14; n= 6, 6, 6, 5, 0, 0, 0 | -87.0 (188.55) | -225.8 (191.16) | -167.7 (159.11) | -125.6 (100.35) |  |  |
  CD4+; Day 17; n= 6, 6, 6, 6, 0, 0, 0 | -85.8 (131.98) | -92.8 (206.08) | -40.7 (247.24) | -79.8 (44.63) |  |  |
  CD4+; Day 21; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD4+; Day 21; n= 6, 5, 6, 6, 0, 0, 0 | -48.5 (102.32) | -209.2 (212.86) | -87.2 (231.76) | -160.0 (54.09) |  |  |
  CD4+; Day 24; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD4+; Day 24; n= 6, 5, 6, 6, 0, 0, 0 | -82.8 (172.46) | -261.4 (119.72) | -126.5 (250.88) | -187.3 (136.51) |  |  |
  CD4+; Day 28; n= 6, 6, 6, 6, 0, 0, 0 | -49.8 (91.84) | -38.5 (210.86) | -206.8 (162.52) | -156.2 (172.35) |  |  |

47. Secondary Outcome: Part 2: Change From Baseline in CD4+ Cells Following Multiple Dose Administration of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for analysis of CD4+ cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

48. Secondary Outcome: Part 1: Change From Baseline in CD8+ Cells Following Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for analysis of CD8+ cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline, Days 2, 3, 5, 8, 11, 14, 17, 21, 24 and 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^6 cells per Liter
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
10^6 cells per Liter
  CD8+; Day 2;n= 6, 6, 6, 6, 0, 0, 0 | -68.3 (63.71) | -41.3 (69.15) | -35.0 (75.52) | -101.2 (102.96) |  |  |
  CD8+; Day 3;n= 6, 6, 6, 6, 0, 0, 0 | -79.5 (103.45) | 22.2 (91.40) | -81.2 (97.61) | -86.0 (84.04) |  |  |
  CD8+: Day 5; n= 6, 6, 5, 6, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0 | 0 | 0
  CD8+: Day 5; n= 6, 6, 5, 6, 0, 0, 0 | -86.8 (85.04) | -60.7 (28.87) | -48.4 (86.25) | -107.5 (110.07) |  |  |
  CD8+; Day 8; n= 6, 6, 6, 6, 0, 0, 0 | -65.7 (57.18) | -26.8 (69.45) | -77.0 (71.26) | -68.7 (56.39) |  |  |
  CD8+; Day 11; n= 6, 6, 6, 6, 0, 0, 0 | -55.0 (52.57) | -52.0 (93.97) | -54.7 (51.45) | -88.5 (61.61) |  |  |
  CD8+; Day 14; n= 6, 6, 6, 5, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0 | 0
  CD8+; Day 14; n= 6, 6, 6, 5, 0, 0, 0 | -81.8 (103.86) | -92.2 (84.57) | -77.5 (45.75) | -96.6 (68.44) |  |  |
  CD8+; Day 17; n= 6, 6, 6, 6, 0, 0, 0 | -50.2 (75.78) | -33.8 (97.41) | 4.7 (84.03) | -83.2 (78.76) |  |  |
  CD8+; Day 21; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD8+; Day 21; n= 6, 5, 6, 6, 0, 0, 0 | -35.8 (35.57) | -74.0 (108.80) | -24.0 (105.96) | -106.5 (90.51) |  |  |
  CD8+; Day 24; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD8+; Day 24; n= 6, 5, 6, 6, 0, 0, 0 | -56.3 (92.88) | -98.0 (99.84) | -53.7 (101.04) | -120.7 (77.79) |  |  |
  CD8+; Day 28; n= 6, 6, 6, 6, 0, 0, 0 | -67.0 (89.66) | 6.3 (128.72) | -127.8 (72.88) | -104.7 (110.66) |  |  |

49. Secondary Outcome: Part 2: Change From Baseline in CD8+ Cells Following Multiple Dose Administration of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for analysis of CD8+ cells. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

50. Secondary Outcome: Part 1: Change From Baseline in CD4+ Cell Median Fluorescence Intensity (MFI) Following Single Dose Administration of GSK3732394
Description: Blood samples were collected at indicated time points for analysis of CD4+ cell MFI. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline, Day 1 (0.5, 1, 2, 4, 8, 12 hours), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 17, 21, 24 and 28
Population: as for outcome 11
Measure: Median (Full Range); unit: Median fluorescence intensity
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Median fluorescence intensity
  CD4+ MFI; Day 1- 0.5 hours; n= 6, 6, 6, 6, 0, 0, 0 | 133.0 [-1358 to 851] | -28.0 [-370 to 810] | 233.0 [-351 to 891] | 742.0 [-703 to 8197] |  |  |
  CD4+ MFI: Day 1- 1 hour; n= 6, 6, 6, 6, 0, 0, 0 | 457.0 [-1293 to 1361] | 109.0 [-1395 to 629] | -48.0 [-757 to 1158] | 693.0 [-276 to 8582] |  |  |
  CD4+ MFI; Day 1- 2 hours; n= 6, 6, 6, 6, 0, 0, 0 | 583.5 [-1482 to 1699] | 197.5 [-1661 to 1008] | 70.0 [-1204 to 1005] | 788.5 [-447 to 6762] |  |  |
  CD4+ MFI; Day 1- 4 hours; n= 6, 6, 6, 6, 0, 0, 0 | 296.0 [-1299 to 627] | 7.5 [-1526 to 1151] | -777.5 [-2204 to 344] | 372.0 [-544 to 9604] |  |  |
  CD4+ MFI; Day 1- 8 hours; n= 6, 6, 6, 6, 0, 0, 0 | -379.5 [-2118 to 1138] | -786.5 [-4129 to 401] | -1870.0 [-4676 to 354] | 747.0 [-1645 to 6519] |  |  |
  CD4+ MFI; Day 1- 12 hours; n= 6, 6, 6, 6, 0, 0, 0 | -358.0 [-2901 to 1622] | -1209.0 [-3343 to 283] | -2788.5 [-3977 to -544] | 536.5 [-1839 to 5954] |  |  |
  CD4+ MFI; Day 2; n= 6, 6, 6, 6, 0, 0, 0 | -241.5 [-1515 to 2496] | -790.5 [-4116 to 1496] | -3486.0 [-5084 to 34] | 354.5 [-1258 to 7124] |  |  |
  CD4+ MFI; Day 3; n= 6, 6, 6, 6, 0, 0, 0 | -351.0 [-2921 to 934] | -839.5 [-4530 to 1258] | -3095.0 [-5157 to -1583] | 1071.5 [227 to 5623] |  |  |
  CD4+ MFI; Day 4; n= 6, 6, 6, 6, 0, 0, 0 | 872.5 [-4236 to 2154] | -427.5 [-4054 to 561] | -2651.5 [-5310 to -602] | 663.5 [-245 to 5169] |  |  |
  CD4+ MFI; Day 5; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD4+ MFI; Day 5; n= 6, 5, 6, 6, 0, 0, 0 | 1665.0 [-1692 to 2659] | -203.0 [-3456 to 1161] | -2374.5 [-5792 to -1434] | 579.0 [-1537 to 6800] |  |  |
  CD4+ MFI; Day 6; n= 6, 6, 6, 6, 0, 0, 0 | 769.5 [-3208 to 3195] | 268.0 [-2048 to 778] | -1807.0 [-4678 to -266] | 1023.5 [-267 to 7103] |  |  |
  CD4+ MFI: Day 7; n= 6, 6, 6, 6, 0, 0, 0 | 1561.0 [-2616 to 2376] | -284.0 [-2308 to 959] | -1129.0 [-3437 to 1044] | 613.0 [-458 to 6433] |  |  |
  CD4+ MFI: Day 8; n= 6, 6, 6, 6, 0, 0, 0 | 1885.5 [-1756 to 2598] | 334.0 [-1755 to 1976] | -580.0 [-3244 to 1397] | 1210.0 [635 to 6949] |  |  |
  CD4+ MFI; Day 9; n= 6, 6, 6, 6, 0, 0, 0 | 1435.5 [-1518 to 2760] | 975.0 [-711 to 1890] | -352.0 [-2295 to 1488] | 1652.5 [-128 to 7726] |  |  |
  CD4+ MFI; Day 10; n= 6, 6, 6, 6, 0, 0, 0 | 1942.5 [-543 to 2610] | 647.5 [-1903 to 2727] | -257.5 [-2762 to 1577] | 1907.0 [-919 to 7195] |  |  |
  CD4+ MFI; Day 11; n= 6, 6, 6, 6, 0, 0, 0 | 2120.5 [-521 to 2678] | 1237.5 [-423 to 2429] | 149.5 [-1436 to 2095] | 1599.0 [404 to 8376] |  |  |
  CD4+ MFI; Day 12; n= 5, 6, 6, 6, 0, 0, 0: number analyzed (Participants) | 5 | 6 | 6 | 6 | 0 | 0 | 0
  CD4+ MFI; Day 12; n= 5, 6, 6, 6, 0, 0, 0 | 1212.0 [-602 to 2770] | 1160.0 [-622 to 1801] | -93.0 [-1471 to 1366] | 1295.0 [-198 to 9007] |  |  |
  CD4+ MFI; Day 13; n= 6, 6, 6, 6, 0, 0, 0 | 1705.5 [-404 to 2996] | 677.5 [-351 to 2137] | 254.5 [-987 to 1378] | 1100.5 [-1294 to 9386] |  |  |
  CD4+ MFI; Day 14; n= 6, 6, 6, 5, 0, 0, 0: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0 | 0
  CD4+ MFI; Day 14; n= 6, 6, 6, 5, 0, 0, 0 | 1760.5 [-2003 to 2297] | 385.5 [-756 to 1882] | 9.5 [-608 to 1438] | 2107.0 [-40 to 6924] |  |  |
  CD4+ MFI; Day 17; n= 6, 6, 6, 6, 0, 0, 0 | 1258.5 [-457 to 2372] | 1024.0 [-606 to 3369] | 809.0 [-554 to 1315] | 391.5 [-926 to 7300] |  |  |
  CD4+ MFI; Day 21;n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD4+ MFI; Day 21;n= 6, 5, 6, 6, 0, 0, 0 | 1663.0 [-287 to 2310] | 955.0 [501 to 1863] | 475.0 [-815 to 1325] | 1247.5 [-654 to 7916] |  |  |
  CD4+ MFI: Day 24; n= 6, 5, 6, 6, 0, 0, 0: number analyzed (Participants) | 6 | 5 | 6 | 6 | 0 | 0 | 0
  CD4+ MFI: Day 24; n= 6, 5, 6, 6, 0, 0, 0 | 1783.5 [-2130 to 2773] | 1382.0 [408 to 2947] | 1039.0 [-542 to 1545] | 1349.5 [200 to 7002] |  |  |
  CD4+ MFI: Day 28; n= 6, 6, 6, 6, 0, 0, 0 | 1193.0 [-731 to 2674] | 1094.5 [-537 to 1689] | 911.0 [-453 to 1611] | 1190.5 [285 to 7860] |  |  |

51. Secondary Outcome: Part 2: Change From Baseline in CD4+ Cell MFI Following Multiple Dose Administration of GSK3732394
Description: Blood samples were planned to be collected at indicated time points for analysis of CD4+ cell MFI. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

52. Secondary Outcome: Part 1: Number of Participants With Anti-GSK3732394 Antibodies on Day 28
Description: Serum samples were collected to analyze antibodies against GSK3732394. The presence of anti-GSK3732394 antibodies was determined in serum samples using a validated bioanalytical method, which included a screening assay, confirmation assay and titer analysis. Positive samples were further characterized with additional assays to determine the specificity of the anti-GSK3732394 antibodies. Number of participants with presence of anti-GSK3732394 antibodies are presented.
Time Frame: Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0
Participants | 6 | 6 | 6 | 1 |  |  |

53. Secondary Outcome: Part 2: Number of Participants With Anti-GSK3732394 Antibodies
Description: Serum samples were planned to be collected to analyze antibodies against GSK3732394.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

54. Secondary Outcome: Part 1: Titer of Anti-drug Antibodies (ADAs) Against GSK3732394 on Day 28
Description: Serum samples were collected to analyze the titers of antibodies against GSK3732394. The presence of anti-GSK3732394 antibodies was determined in serum samples using a validated bioanalytical method, which included a screening assay, confirmation assay and titer analysis. Positive samples were further characterized with additional assays to determine the specificity of the anti-GSK3732394 antibodies. Positive samples were titrated to obtain the titers of antibodies.
Time Frame: Day 28
Population: Safety Population. Data was not collected for Cohort 4 to 6, as the study was terminated after Part 1-Cohort 3 and hence no participants were enrolled. Only those participants with data available at the specified data points were analyzed. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Median (Full Range); unit: Titer
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394
Number analyzed (Participants) | 6 | 6 | 6 | 1 | 0 | 0 | 0
Titer | 2000.0 [160 to 32000] | 240.0 [40 to 16000] | 8500.0 [320 to 256000] | 40.0 [40 to 40] |  |  |

55. Secondary Outcome: Part 2: Titer of ADAs Against GSK3732394
Description: Serum samples were planned to be collected to analyze the titers of antibodies against GSK3732394.
Time Frame: Up to Day 49
Population: as for outcome 2
Arm/Group | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from start of study intervention (Day 1) up to Day 28.
Description: Safety Population consisted of all participants who received at least 1 dose of study treatment. Data is presented for Part 1- Cohorts 1 to 3. Non-SAEs and SAEs were not collected for Part 1 (Cohorts 4 to 6) and Part 2 as the study was terminated after Part 1-Cohort 3.
Arm/Group | Part 1- Cohort 1: GSK3732394 10 mg | Part 1- Cohort 2: GSK3732394 20 mg | Part 1- Cohort 3: GSK3732394 80 mg | Part 1- Placebo | Part 1- Cohort 4: GSK3732394 | Part 1- Cohort 5: GSK3732394 | Part 1- Cohort 6: GSK3732394 | Part 2- Cohort 1: GSK3732394 | Part 2- Cohort 2: GSK3732394 | Part 2- Cohort 3: GSK3732394 | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 4/6 | 2/6 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1- Cohort 1: GSK3732394 10 mg (N=6) | Part 1- Cohort 2: GSK3732394 20 mg (N=6) | Part 1- Cohort 3: GSK3732394 80 mg (N=6) | Part 1- Placebo (N=6) | Part 1- Cohort 4: GSK3732394 (N=0) | Part 1- Cohort 5: GSK3732394 (N=0) | Part 1- Cohort 6: GSK3732394 (N=0) | Part 2- Cohort 1: GSK3732394 (N=0) | Part 2- Cohort 2: GSK3732394 (N=0) | Part 2- Cohort 3: GSK3732394 (N=0) | Part 2: Placebo (N=0)
Injection site hypersensitivity (General disorders) | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03984812/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT03984812/SAP_001.pdf